CLINICAL TRIAL: NCT01259830
Title: A Double-blind, Randomized, Placebo Controlled Study to Evaluate the Effectiveness of Etoricoxib as an Additive Analgesic to Epidural Analgesia in Colon or Rectal Fast-track Surgery
Brief Title: Effectiveness of Etoricoxib as an Additive Analgesic to Epidural Analgesia in Colon or Rectal Fast-track Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Claudia Spies (Other)
Responsible Party: Sponsor-Investigator, Claudia Spies, Prof. MD, Director of the Dept. of Anesthesiology and Intensive Care Medicine, CVK, CCM, Charite University, Berlin, Germany, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Etoricoxib-fast-track
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Post-operative Pain
Keywords: fast-track; colon or rectal surgery; pain relief
MeSH Terms: conditions — Pain, Postoperative | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arcoxia® 120 mg (Experimental)
  Interventions: Drug: Arcoxia®120 mg
- Sugar pill (Placebo Comparator)
  Interventions: Drug: P Tablet White Lichtenstein

INTERVENTIONS:
Drug: Arcoxia®120 mg — Arcoxia® over encapsulated 120 mg; Perioperatively 6 days 1 tablet (Arcoxia® 120 mg) for oral use
  Other Names: Etoricoxib
  Arms: Arcoxia® 120 mg
Drug: P Tablet White Lichtenstein — P Tablet White Lichtenstein over encapsulated; Perioperatively 6 days 1 tablet for oral use
  Arms: Sugar pill

SUMMARY:
Post-operative pain after laparoscopic colon and rectal surgery in fast-track design.

A fast-track program is an evidence-based, multimodal approach for patients undergoing surgery to reduce perioperative morbidity, hospital stay and cost and to increase patient centered well-being. Optimized pain relief is a core component of any fast-track regimen.

In this context epidural analgesia has become the standard of care for early postoperative pain therapy.

However, it is debated whether non-opioid analgesics should be given as adjuncts when epidural analgesia is already present.

The purpose of this study is to demonstrate that the administration of etoricoxib 120mg additionally to the clinical routine therapy (epidural catheter) reduces the post-operative pain level during movement after laparoscopic colon surgery in the fast-track design.

DETAILED DESCRIPTION:
A fast-track program is an evidence-based, multimodal approach for patients undergoing surgery to reduce perioperative morbidity, hospital stay and cost and to increase patient centered well-being. Particularly in visceral surgery of the colon it is gaining widespread acceptance (Schwenk 2009). Optimized pain relief is a core component of any fast-track regimen (Kehlet and Wilmore 2008). In this context epidural analgesia has become the standard of care for early postoperative pain therapy (Hasenberg 2009), providing superior pain relief compared to parenteral opioids (Block 2001).

However, it is debated whether non-opioid analgesics should be given as adjuncts when epidural analgesia is already present. Some studies have found reduced pain using NSAID as adjunct (Scott 1994), leading to a positive recommendation in the German guidelines for postoperative pain therapy (S3-Leitlinie). However, other studies (Mogensen 1992) have not found an effect of non-opioids in addition to epidural analgesia. Further studies are also needed to assess whether nonopioid adjuncts can facilitate the change from epidural to systemic analgesia (typically on the 2nd or 3rd postoperative day) and reduce opioid consumption during the days after catheter removal.

Fast-track surgery is a multi-model process, and every step in this process needs to be fine-tuned to yield best results (Langelotz 2005). Until now studies have compared only groups with either epidural or systemic analgesia, but for optimal recovery a sequential approach with a combination of both is probably a better choice. A typical multimodal analgesia regimen after removal of an epidural at our institution consists of acetaminophen and ibuprofen. Opioids are avoided if possible, but are added if needed. An improved non-opioid analgesia regimen is a sought-after goal in this fast-track-phase. The study is controlled in terms of the type of surgery (laparoscopic colon and rectal surgery) and all factors of the multimodal analgesia treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or over
* written informed consent
* no inclusion in other medical studies according to the AMG (German drug law) during the study period
* realization of colon or rectal surgery in the fast track design after clinical standards including an epidural catheter

Exclusion Criteria:

* ASA status IV-V
* allergy against etoricoxib, other components or other NSAID
* coronary heart disease
* heart insufficiency NYHA II-IV
* cerebrovascular disease
* peripheral arterial occlusive disease
* untreated arterial hypertonus
* active peptic ulcera or active gastrointestinal bleeding
* minor to severe liver dysfunction (beginning from Child - Plugh - Classification A)
* kidney insufficiency
* inflammatory bowel disease
* pregnancy (positive hCG laboratory test) or lactation
* Women of child-bearing potential who are not using a highly effective contraception method with a pearl-index < 1 during study participation and for at least 3 consecutive months after study inclusion.
* placement in an institution on order of an official authority
* missing consent for saving and passing on pseudonymous data
* hereditary galactose-intolerance, lactase deficit, glucose-galactose-malabsorption
* no correct epidural catheter placement within 48 h after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Primary end point of the study is the average pain level (scale 0-10) in the area of surgery during movement (walking a fixed number of steps) under active epidural analgesia, at the third day following laparoscopic colon or rectal surgery. | Third postoperative day
  To demonstrate that the administration of etoricoxib 120mg additionally to the clinical routine therapy (epidural catheter) reduces the post-operative pain level during movement at the third day after laparoscopic colon or rectal surgery in the fast-track design.

SECONDARY OUTCOMES:
Post-operative pain level during movement in the first 2 days after laparoscopic colon or rectal surgery. | In the first 2 days after laparoscopic colon or rectal surgery
Post-operative pain level during rest in the first 2 days after laparoscopic colon or rectal surgery. | In the first 2 days after laparoscopic colon or rectal surgery
Post-operative pain level during rest and movement from the third (one day after epidural catheter removal) until the fifth day after laparoscopic colon or rectal surgery | In the first three days after epidural catheter removal
Incidence of pain events and the average pain intensity in body parts outside of the area of operations. | In the first three days after epidural catheter removal
Incidence of new organ dysfunctions | In the first nine days after laparoscopic colon or rectal surgery
  Organ dysfunctions (cardiovascular, gastrointestinal, renal, respiratory, cognitive, infective)
Postoperative LOS | Period of hospital stay, an exspected average of seven days
Patients level of satisfaction | In the first five days after laparoscopic colon or rectal surgery
Incidence of side effects | In the first nine days after laparoscopic colon or rectal surgery
  Side effects by IMP
Postoperative intensive care unit stay | Period of intensive care unit stay, an exspected average of one day
Amount and frequency of intake of rescue medication | In the first five days after laparoscopic colon or rectal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Dept. of Anesthesiology and Intensive Care, Charité, Universitätsmedizin Berlin
Locations (4):
- Germany (4):
  - St. Hedwig Kliniken Berlin GmbH, Department of Anesthesiology and Intensive Care Medicine, Berlin, State of Berlin
  - Department of Anesthesiology, Sana-Klinikum Lichtenberg, Oskar-Ziethen-Krankenhaus, Berlin, State of Berlin
  - Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum/Campus Charité Mitte, Charité Universitätsmedizin, Berlin, State of Berlin
  - Department of Anesthesiology, Johannes Wesling Klinikum Minden Mühlenkreiskliniken (AöR), Minden